CLINICAL TRIAL: NCT07030699
Title: Epcoritamab With Lenalidomide and Tafasitamab in Patients With Relapsed/Refractory (R/R) Diffuse Large B Cell Lymphoma (DLBCL)
Brief Title: A Study of Epcoritamab With Lenalidomide and Tafasitamab in People With Diffuse Large B Cell Lymphoma
Acronym: ECLAT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Genmab (Industry); Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-070
Record Dates: First submitted 2025-06-12; First posted 2025-06-22 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Lymphoma
Keywords: Large B cell lymphoma; Transformed indolent lymphoma; Primary mediastinal B cell lymphoma; High grade B cell lymphoma; Follicular lymphoma grade 3B; Epcoritamab; Lenalidomide; Tafasitamab; 25-070
MeSH Terms: conditions — Lymphoma | interventions — Lenalidomide; tafasitamab

STUDY DESIGN:
Intervention Model Description: This is a phase 2, open label, single arm, single institution study.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Epcoritamab with Lenalidomide and Tafasitamab (Experimental): Epcoritamab: Subcutaneous, once weekly in cycles 1-3; every 4 weeks cycles 4-12. Tafasitamab: Intravenous, once weekly during cycles 1-3, then every 2 weeks during cycle 4-12. Lenalidomide: Oral, daily on days 1-21 of a 28-day cycle.
  Interventions: Drug: Epcoritamab; Drug: Lenalidomide; Drug: Tafasitamab

INTERVENTIONS:
Drug: Epcoritamab — Subcutaneous, once weekly in cycles 1-3; every 4 weeks cycles 4-12
Drug: Lenalidomide — Oral, daily on days 1-21 of a 28-day cycle
Drug: Tafasitamab — Intravenous, once weekly during cycles 1-3, then every 2 weeks during cycle 4-12

SUMMARY:
The researchers are doing this study to find out whether the combination of epcoritamab with tafasitamab and lenalidomide is a safe and effective treatment for relapsed or refractory DLBCL. This is the first time the combination of drugs is being tested.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Pathologically confirmed diffuse large B cell lymphoma, transformed indolent lymphoma, primary mediastinal B cell lymphoma, high grade B cell lymphoma, follicular lymphoma grade 3B
* Subjects must have histologically confirmed CD20+ lymphoma as documented in the most recent representative pathology report.
* Presence of CD19 is not required to be confirmed (except if patients have received anti-CD19 therapy in the past). Patients treated with prior anti-CD19 therapy must have confirmation of CD19 expression in a biopsy done after progression on the last CD19 directed therapy.
* At least 2 prior lines of systemic therapy including CART or ASCT (up to 4 prior lines of therapy allowed). Note that bridging therapy prior to ASCT or CART will be counted as a separate line of therapy)
* At least one prior line of systemic therapy for patients ineligible for ASCT/CART or patients unwilling to undergo CAR-T/ASCT for logistic or other reasons (up to 4 prior lines of therapy allowed)
* Have radiologically measurable lymphadenopathy or extranodal involvement.
* Eastern Cooperative Oncology Group performance status (PS) ≤ 2 (ECOG >2 can be enrolled if PS compromised from lymphoma e.g. spinal cord compression and expected to improve rapidly with therapy)
* Must have adequate organ and marrow status Hemoglobin ≥8 g/dL (red blood cell transfusions are allowed)

  * Absolute neutrophil count (ANC) ≥1,000/mm^3 or ≥500/mm^3 if due to disease involvement in the bone marrow (G-CSF use is allowed).
  * Platelet count ≥75,000 cells/mm^3 or ≥50,000/mm^3 if due to disease involvement in the bone marrow (platelets transfusions are allowed)
  * Estimated Creatinine Clearance (CrCl) ≥40 mL/min (Cockcroft-Gault formula or other institutional standard methods)
  * Serum aspartate transaminase (AST) or alanine transaminase (ALT) ≤2.5 x upper limit of normal (ULN)
  * Direct bilirubin ≤ 2 x ULN (≤3 if due to Gilbert's syndrome or liver involvement by the lymphoma)
* Negative HIV test at screening, with the following exception: Individuals with a positive HIV test at screening are eligible provided, prior to enrollment, they are stable on antiretroviral therapy for at least 1 year, have a CD4 count ≥ 200/μL, and have an undetectable viral load.
* Signed Informed Consent Form(s)
* Ability to comply with all the study-related procedures, in the investigator's judgement
* Subject is willing to take aspirin prophylaxis (subjects with low or intermediate risk for thromboembolism) or prophylactic anticoagulant (if high risk for a thromboembolic event)
* Contraception requirements

  * Patient is willing to adhere to pregnancy risk minimization plan associated with lenalidomide treatment.
  * For all females of child-bearing potential; a negative serum pregnancy test (beta-hCG) at the Screening Visit and a negative serum or urine pregnancy test at baseline prior to the first dose of study drug.
  * Female subjects of childbearing potential must practice at least 2 protocol-specified methods of birth control, that are effective from 30 days prior to treatment through at least 12 months after the last dose of study drug.
  * Female subjects of non-childbearing potential do not need to use birth control.
  * Female who is not pregnant, breastfeeding, donating eggs (ova, oocytes), or considering
  * becoming pregnant during the study or for 12 months after the last dose of study drug.
  * If male, and subject is sexually active with female partner(s) of childbearing potential, he must agree, from 30 days prior to treatment initiation through 12 months after the last dose of study drug, to practice the protocol-specified contraception.
  * Male who is not considering fathering a child or donating sperm during the study or for 12 months after the last dose of study drug.
* COVID19 eligibility criteria: Patient should have no known active severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection. If a patient has signs/symptoms suggestive of SARS-CoV-2 infection or have had recent known exposure to someone with SARS-CoV-2 infection, the subject must have a negative molecular (e.g., PCR) test, or 2 negative antigen test results at least 24 hours apart, to rule out SARS-CoV-2 infection. Note: SARS-CoV-2 diagnostic tests should be applied following local requirements/recommendations.
* Subjects who do not meet SARS-CoV-2 infection eligibility criteria must be screen failed and may only rescreen after they meet the following SARS-CoV-2 infection viral clearance criteria:

  * No signs/symptoms suggestive of active SARS-CoV-2 infection
  * Negative molecular (e.g., PCR) result or 2 negative antigen test results at least 24 hours apart

Exclusion Criteria:

* Prior CD3/CD20 BiAb based therapy with the following exceptions:

  * Patients who received prior CD3/CD20 BiAb as part of frontline therapy for DLBCL and were in remission for at least 1 year post frontline therapy are allowed
  * Patients who received prior CD3/CD20 BiAb as part of bridging therapy prior to CAR-T cell therapy without documentation of refractory/progressive disease on CD/CD30 BiAb are allowed
  * Patients who received prior CD3/CD20 BiAb and were in remission for at least 6 months after last dose of drug are allowed
* Prior tafasitamab and/or lenalidomide therapy for lymphoma

  * Patients who received prior tafasitamab and/or lenalidomide as part of frontline therapy for DLBCL and were in remission for at least 1 year post frontline therapy are allowed
  * Patient who received prior lenalidomide without evidence of intolerance or progression on drug are allowed
* Active CNS involvement (previously treated CNS lymphoma is permissible)
* Active secondary malignancy

  * Patients who have a concurrent malignancy that is clinically stable and does not require tumor-directed treatment is allowed e.g., low grade prostate cancer under surveillance
  * Patients with a previously treated malignancy should be eligible to participate if all treatment of that malignancy was completed at least 2 years before registration and the patient has no evidence of disease.
  * Other cases of active concurrent malignancies may be considered on a case-by-case basis if benefit outweighs risk after discussion with PI
* Uncontrolled HIV or active HBV or HCV infection (controlled HIV with undetectable viral load, previously treated HBV and HCV are allowed if HBV DNA and HCV RNA are negative respectively, HBcAb positive with HBsAg negative disease is permitted if patient is willing to take entecavir prophylaxis)
* Known active or latent tuberculosis
* Prior solid organ transplantation
* Prior allogeneic stem cell transplantation
* Uncontrolled active systemic infection
* Major surgery within 4 weeks of the first dose of study drug (exceptions may be allowed after discussion with PI if patient has fully recovered from procedure and anti-lymphoma therapy is urgently needed)
* Known clinically significant cardiovascular disease, including:

  * Onset of unstable angina pectoris within 6 months of signing ICF
  * Acute myocardial infarction within 6 months of signing ICF
  * Uncontrolled congestive heart failure (grade III or IV as classified by the New York Heart Association)
  * Stroke or intracranial hemorrhage within 6 months prior to signing ICF In case of any other history of major cardiovascular disease, a cardiology consult is required within 60 days of enrollment
* Any life-threatening illness, medical condition, or organ system dysfunction that, in the investigator's opinion, could compromise the subject's safety or risk study outcomes
* Vaccination with live vaccines within 28 days prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-08-13 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
best complete response rate (CRR) | 2 years
  CR rate based on PET scan, as determined by the investigator according to the Lugano Response Criteria for Malignant Lymphoma (hereafter referred to as the 2014 Lugano Response Criteria)

CONTACTS AND LOCATIONS:
Overall Officials: Pallawi Torka, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center Suffolk - Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org